CLINICAL TRIAL: NCT06703242
Title: Non-randomized Controlled Pilot Study of a Health Promotion Program for Mothers of Children in the Ultra-orthodox Community: Examining Feasibility
Brief Title: Pilot Study on a Health Promotion Intervention for Ultra-Orthodox Mothers of Children With ADHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adina Maeir (Other)
Collaborators: Monash University (Other)
Responsible Party: Sponsor-Investigator, Adina Maeir, Professor, Hebrew University of Jerusalem
Organization: Hebrew University of Jerusalem (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 30012024
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Attention Deficit Disorder With Hyperactivity (ADHD)
Keywords: Mothering a child with ADHD; Maternal psychological health; Ultra-orthodox
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: Mothers in the control group will receive the intervention right after the completion of the intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Health promotion intervention group (Other): A one time six-session weekly intervention group for mothers of children with ADHD in the ultra-orthodox community.
  Interventions: Other: Health promotion for mothers of children with ADHD in the ultra-orthodox community

INTERVENTIONS:
Other: Health promotion for mothers of children with ADHD in the ultra-orthodox community — The intervention will consist of 3 modules with six sessions. Mothers will gain knowledge in topics related to understanding the ADHD health condition and its biological origins, optimal and recommended treatment options, school management techniques, and the importance of taking care of their own health.

SUMMARY:
The goal of this study is to evaluate the feasibility and effectiveness of a health promotion intervention for Ultra-Orthodox Jewish mothers of children with ADHD.

This study will examine the impact of a culturally tailored group-based intervention aimed at reducing stress, enhancing health, and improving the well-being of mothers.

The main questions this study aims to answer are:

1. Is the intervention feasible for mothers to participate?
2. Does the intervention improve maternal knowledge about ADHD and reduce stigma?
3. Does it help reduce maternal stress and enhance self-care practices?

Participants include:

Mothers: Ultra-Orthodox Jewish mothers with a child (ages 6-12) diagnosed with ADHD and no other major health conditions in the family (other than ADHD).

Educators: School educators with at least 5 years of experience teaching children with ADHD in the Ultra-Orthodox community.

What participation involves:

Mothers will attend six weekly teletherapy group sessions, with 6-8 mothers per group. They will complete questionnaires before and after the intervention (approximately 30 minutes each) and participate in a 90-minute remote focus group to provide feedback on the program.

Educators will attend a single teletherapy group session (90 minutes) during the program (session 5) and participate in a 90-minute remote interview to provide feedback on the program.

DETAILED DESCRIPTION:
After providing informed consent, mothers will complete questionnaires which will take approximately 30 minutes before beginning the program. Mothers will then be assigned non-randomly to the intervention or control group. Mothers assigned to the control group will receive the intervention after the completion of the first intervention group (delayed).

The six sessions of the intervention will be teletherapy and each session will be one and a half hours in length. Each group will consist of 6-8 mothers per group.

Inclusion criteria included mothers who identify as ultra-orthodox Jewish, have a child between the ages of 6-12 years old who have been diagnosed with ADHD by a licensed medical professional, and who do not have any other medical diagnosis.

The topics discussed in the intervention will include: Awareness/knowledge regarding ADHD and its biological origins, Identifying resources and optimal treatment for ADHD for the child and the mother, Strategies for child ADHD management in the school, and the legitimacy and importance of maternal self-care.

ELIGIBILITY:
Inclusion Criteria:

* mothers of children with ADHD aged 6- 12 years old
* Mothers who identify as ultra-orthodox Jews
* Child diagnosis was by a licensed medical professional

Exclusion Criteria:

* Child medical diagnosis other than ADHD

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Change in maternal ADHD Knowledge as measured by the ADHD Knowledge Questionnaire (Bussing, 2014) | from enrollment until the end of the six week sessions of the intervention
  The summary knowledge score is composed of the sum of 5 variables:
  1. Ever heard of ADHD (no =0; yes= 1)
  2. Recency of information (0= heard months to years ago or never; 1= heard days to weeks ago)
  3. Self-rated knowledge amount (0= knows little to nothing; 1 =knows some or a lot)
  4. Number of information sources used (0= none or one; 1 = two or more sources cited)
  5. Attribution of ADHD to sugar in the diet (0= probably or definitely true; 1 =probably or definitely false).
  Knowledge scores can range from 0 to 5 ('0' indicating the least amount of knowledge), and were normally distributed (mean =2.6, SD =1.6, median =3)
Change in maternal ADHD stigma as measured by the ADHD Stigma Scale | from enrollment until the end of the six week sessions of the intervention
  The questions ask about some of the experiences, feelings, and opinions people with ADHD might have and how they are treated. Each item is rated on a 4-point Likert scale (1=strongly disagree; 2=disagree; 3-agree; 4=strongly agree), with higher scores indicating higher stigma perceptions.
  The overall stigma score is composed of the sum of all 26 items
Change in maternal stress as measured by the Parental Stress Items | from enrollment until the end of the six week sessions of the intervention
  Parenting Stress Items measures parental stress, by asking parents to consider how "tense" or "frustrated" they feel about parenting their children. Includes 11 items scored on a four-point scale (1¼not at all to 4¼very much so), yielding scores ranging from 11-44, with higher scores indicating greater levels of parenting stress.
Change in maternal participation in health promoting activities as measured by the Health Promoting Activities Scale | from enrollment until the end of the six week sessions of the intervention
  Health Promoting Activities Scale (HPAS) is an eight-item measure that assesses frequency of participation in social, emotional, physical, and spiritual leisure activities on a seven-point scale (1=never to 7=once or more every day). Scores range from 8 to 56, with higher scores indicating more frequent participation

CONTACTS AND LOCATIONS:
Overall Officials: Adina Maeir, PhD, Principal Investigator — Hebrew University
Locations (1):
- Hebrew University, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
Study protocol Statistical analysis plan Informed consent form All IPD that are part of the results section in a publication
Supporting Information: Study Protocol, ICF
Time Frame: The study protocol and informed consent form are already available. The statistical analysis plan will be available within 6 months of publication.
Access Criteria: De-identified individual participant data (IPD), including questionnaire and statistical analysis results, will be shared upon reasonable request for research purposes. Access will be granted to qualified researchers affiliated with academic, healthcare, or research institutions for analyses advancing knowledge of ADHD interventions, maternal health, or culturally tailored health promotion programs.
  Requests must be submitted in writing to the principal investigator (PI) and include:
  A summary of the request's purpose. Institutional affiliation and researcher qualifications. A data use agreement ensuring confidentiality and ethical compliance. The PI and a review panel will evaluate requests based on scientific validity and alignment with study goals. Approved data will be shared via secure methods, such as encrypted file-sharing platforms, in compliance with privacy regulations. Data will be available 6 months after publication and remain accessible for 2 years.

REFERENCES:
- [Background] Budman JR, Maeir A. Development of a psychological health promotion intervention for ultra-orthodox Jewish mothers of children with ADHD using the intervention mapping protocol. BMC Public Health. 2024 Feb 29;24(1):645. doi: 10.1186/s12889-024-18126-4. PMID 38424536
- [Background] Budman JR, Fogel-Grinvald H, Maeir A. Psychological Health and Quality of Life among Ultra-orthodox Mothers of Children with Attention Deficit Hyperactivity Disorder: Impact of Occupational Experiences. Phys Occup Ther Pediatr. 2023;43(6):697-712. doi: 10.1080/01942638.2023.2188077. Epub 2023 Mar 15. PMID 36922732
- [Background] Budman J, Maeir A. Mothering a Child with ADHD in the Ultra-Orthodox Community. Int J Environ Res Public Health. 2022 Nov 4;19(21):14483. doi: 10.3390/ijerph192114483. PMID 36361375
- [Background] Bourke-Taylor H, Lalor A, Farnworth L, Pallant JF. Further validation of the Health Promoting Activities Scale with mothers of typically developing children. Aust Occup Ther J. 2014 Oct;61(5):308-15. doi: 10.1111/1440-1630.12137. Epub 2014 Sep 9. PMID 25201148
- [Background] Bussing R, Zima BT, Mason DM, Meyer JM, White K, Garvan CW. ADHD knowledge, perceptions, and information sources: perspectives from a community sample of adolescents and their parents. J Adolesc Health. 2012 Dec;51(6):593-600. doi: 10.1016/j.jadohealth.2012.03.004. Epub 2012 Apr 17. PMID 23174470
- [Background] Kellison I, Bussing R, Bell L, Garvan C. Assessment of stigma associated with attention-deficit hyperactivity disorder: psychometric evaluation of the ADHD stigma questionnaire. Psychiatry Res. 2010 Jul 30;178(2):363-9. doi: 10.1016/j.psychres.2009.04.022. Epub 2010 May 23. PMID 20580842
- [Background] Pearlin LI, Schooler C. The structure of coping. J Health Soc Behav. 1978 Mar;19(1):2-21. No abstract available. PMID 649936

DOCUMENTS (2):
  • Study Protocol (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT06703242/Prot_000.pdf
  • Informed Consent Form (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/42/NCT06703242/ICF_001.pdf